CLINICAL TRIAL: NCT01165190
Title: Effect of Pioglitazone on Mitochondrial Function in Muscle and Adipose Tissue in Humans
Acronym: PIO
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-012A
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, and adipose tissue will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pioglitazone group
  Interventions: Other: pioglitazone

INTERVENTIONS:
Other: pioglitazone

SUMMARY:
Mitochondrial dysfunction in skeletal muscle results in decreased muscle fatty acid oxidation, leading to conversion of fatty acids into triglycerides and its accumulation inside the muscle tissue. Moreover, in adipose tissue mitochondrial dysfunction results in decreased fatty acid oxidation and triglyceride synthesis, leading to increased circulating fatty acid concentrations, which in turn also leads to lipid accumulation inside muscle tissue. Lipid accumulation inside muscle tissue interferes with the insulin signaling pathway and causes insulin resistance. Mitochondrial dysfunction in both tissues has therefore been proposed to play an important role in insulin resistance in humans.

Pioglitazone, a thiazolidinedione, is an FDA approved medication for the treatment of type 2 diabetes. It improves muscle insulin sensitivity at least in part by lowering intramuscular lipid concentrations but the mechanism by which this occurs is unclear. In the present study, we shall therefore test the hypothesis that pioglitazone improves mitochondrial function in muscle and adipose tissue in humans who are insulin resistant.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
3. Subjects must range in age from 18-65.
4. Subjects must have the following laboratory values:

   * 2-hour OGTT plasma glucose 140-250 mg/dl
   * Hematocrit ≥ 35 vol%
   * Serum creatinine ≤ 1.6 mg/dl
   * AST (SGOT) < 2.5 times upper limit of normal
   * ALT (SGPT) < 2.5 times upper limit of normal
   * PT, PTT within the normal range

Exclusion Criteria:

1. Subjects must not be receiving any medications with known effects on glucose tolerance unless the subject has been on stable dose of such agents for the past three months before entry into the study. Subjects taking systemic glucocorticoids will be excluded. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months.
2. History of clinically significant heart disease, including ischemic heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG) and congestive heart failure
3. History of peripheral vascular disease (history of claudication)
4. History of pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation).
5. History of peripheral edema
6. Uncontrolled hypertension with systolic BP>160 mmHg, diastolic BP>100 mmHg
7. Resting heart rate >100 beats/min
8. Autonomic neuropathy
9. Heavy alcohol consumption (> 2 drinks/day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women, ages 18-65, any ethnicity.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Distribution of adipocyte mitochondria | 3 months

SECONDARY OUTCOMES:
number of adipocyte proteins | 3 months
number of mitochondrial proteins | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Research Unit, Tempe, Arizona
  - Tempe, Arizona

REFERENCES:
- [Result] Xie X, Sinha S, Yi Z, Langlais PR, Madan M, Bowen BP, Willis W, Meyer C. Role of adipocyte mitochondria in inflammation, lipemia and insulin sensitivity in humans: effects of pioglitazone treatment. Int J Obes (Lond). 2017 Aug 14:10.1038/ijo.2017.192. doi: 10.1038/ijo.2017.192. Online ahead of print. PMID 29087390